CLINICAL TRIAL: NCT04612582
Title: A Comparative Study of Bortezomib-Thalidomide-Dexamethason and Bortezomib-Cyclophosphamide-Dexamethason in the Treatment of Monoclonal Immunoglobulin Light Chain Amyloidosis: A Prospective Randomized Controlled Trial（BTD-CHINA-TRIAL）
Brief Title: Comparison of BTD and BCD Based Regimens in the Treatment of AL Amyloidosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WJWang001
Record Dates: First submitted 2020-06-15; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-04

CONDITIONS: Immunoglobulin Light-Chain Amyloidosis
Keywords: AL Amyloidosis; Bortezomib; cyclophosphamide; thalidomide; randomized controlled trial; prognosis; Side effect
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — Thalidomide; Bortezomib; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Patients who meet the entry criteria will randomly enter the BTD or BCD treatment group according to the proportion of 1:1. The random code will be generated by computer and the random envelope will be made according to the random code. Treatment group included. Each code has a corresponding random envelope. According to the time sequence of subjects meeting the entry criteria, the random number of subjects will be given from small to large. The corresponding random envelope can only be opened during grouping. If a random number falls off in the middle of use, it can no longer be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group1 (Experimental): Group1 is the AL amyloidosis patients who have bortezomib-thalidomide-dexamethason-based regimens for their treatment.
  Interventions: Drug: Thalidomide
- Group2 (Experimental): Group2 is the AL amyloidosis patients who have bortezomib-cyclophosphamide-dexamethason-based regimens for their treatment.
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Thalidomide — Bortezomib (d 1, 8, 15, 22, 1.3mg /m2, subcutaneous injection); thalidomide (d 1-28 50-100mg, oral); dexamethason (d 1, 2, 8, 9, 15, 16, 22, 23, 20mg, oral/intravenous injection) as a course of treatment, the patients will complete six courses of treatment after entering the group, and the total observation time is one year after the end of treatment.
  Other Names: Bortezomib; Dexamethason
  Arms: Group1
Drug: Cyclophosphamide — Bortezomib (d 1, 8, 15, 22,1.3mg / m2, subcutaneous injection); cyclophosphamide (d 1, 2,900mg / m2, intravenous drip); dexamethason (d 1, 2, 8, 9,15, 16, 22, 23, 20mg, oral/intravenous injection) as a course of treatment, patients will complete six courses of treatment after entering the group, the overall observation time is one year after the end of treatment.
  Other Names: Bortezomib; Dexamethason
  Arms: Group2

SUMMARY:
Research Objective:At present, there is no standard therapeutic regimen for monoclonal immunoglobulin light chain (AL) amyloidosis in the world. To compare the efficacy and safety of the regimens between bortezomib-thalidomide-dexamethasone (BTD) and bortezomib-cyclophosphamide-dexamethasone (BCD) in the treatment of AL amyloidosis, so as to provide more clinical evidence for the standard treatment for the disease.

Research Design:This study was designed as a prospective, randomized and controlled clinical study. Patients who meet the inclusion criteria of this study will be randomized to the BTD scheme group or BCD scheme group.

DETAILED DESCRIPTION:
Object and source:Patients meeting the inclusion criteria of AL amyloidosis are enrolled into the study. Screening failure rate ≤ 30%, follow-up dropout rate ≤ 10%.

Sample size evaluation: The complete remission rate (CR) and the very good partial remission rate (VGPR) were used as statistical indexes for hematology remission rate estimation. Referring to the previous literature, the CR and VGPR of bortezomib-thalidomide-dexamethasone (BTD) is 83%, and CR and VGPR of bortezomib-cyclophosphamide-dexamethasone (BCD) is 43%. The boundary value is 0.1, according to the level of significance level α = 0.05, test efficacy 1 - β = 0.8, using the method of effectiveness test, using pass11 software calculation to estimate the sample size to be included in the group, the expected dropout rate is 20%, the total sample size is 70, 35 in each group.

Observation index:Before and after treatment, physical examination should be carried out every month. The following test should be required. Blood pressure

, blood routine, liver function, electrolyte, 24h urine volume, 24h urine protein quantity, urine protein/creatinine ratio, blood uric acid, serum albumin, urea nitrogen, creatinine, eGFR(estimated Glomerular Filtration Rate), blood lipids, infection index, NT-proBNP (N terminal pro B type natriuretic peptide), TNT(Troponin-T), blood and urine free light chain should be detected respectively.

Quality assurance plan:The study shall be conducted in accordance with the current approved protocol and the July 1996 ICH drug clinical study management code (CPMP/ICH / 135/95) (ICH GCP), the Helsinki declaration, regulations and standard operating procedures.

Plan for missing data:(1)When the subject falls off, the researcher should contact the subject as soon as possible by means of visiting, making an appointment for follow-up, making phone calls, sending letters, etc., asking the reason, making record as much detail as possible.(2)All patients with abscission should be recorded for ITT analysis. There is no need for replacement for exfoliated patients. (3)If a patient withdraws from the study due to anaphylaxis, adverse reactions or ineffective treatment, the investigator shall take corresponding treatment measures according to the actual situation of the subject.

Statistical analysis plan:The main evaluation indexes were hematology CR and VGPR, organ function CR and VGPR. The statistical index of treatment effect is the number of patients who meet the criteria of CR and VGPR. Conclusion: if P > 0.05, H0 hypothesis cannot be rejected according to the test level of single side α = 0.05, that is to say, it cannot be judged that the treatment of light amyloidosis in BTD group is better than that in BCD group; if P ≤ 0.05, it can be considered that the treatment of light amyloidosis in BTD group is better than that in BCD group. The difference between the two groups was analyzed by chi square test or Fisher exact probability test as a secondary evaluation index (the overall survival rate and progression free survival period were observed after one year follow-up after six courses of treatment).The safety analysis set includes all cases entering the study and using at least one dose of the study drug. Chi square test or Fisher exact probability test were used to analyze the incidence of adverse events in the two groups. Chi square test or McNemar test were used to analyze the change of abnormal rate of laboratory indexes from baseline.

ELIGIBILITY:
Inclusion Criteria:

1.Signed the written informed consent; 2.18 years old ≤ age ≤ 80 years old, no restriction on gender; 3.AL amyloidosis was confirmed by pathological biopsy in the accumulated system or organ (kidney, heart, liver, skin), and excluded other secondary factors; 4.The proliferation of monoclonal plasma cells was confirmed by fixed electrophoresis of bone marrow or blood/urine.

Exclusion Criteria:

1. Pathological biopsy showed non-AL amyloidosis;
2. Abnormal proliferation of plasma cells reached the standard of multiple myeloma；
3. Other hematological system tumors;
4. Cushing's syndrome;
5. Active hepatitis;

5.Pregnant or lactating women;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Hematologic Response | 1 year
  According to the criteria of hematologic response of AL amyloidosis.

SECONDARY OUTCOMES:
Organ Response | 1 year
  According to the criteria of organ response of AL amyloidosis.

CONTACTS AND LOCATIONS:
Overall Officials: Wenjian Wang, PhD, Study Chair — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People'S Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang XH, Liu ZH. The Clinical Presentation and Management of Systemic Light-Chain Amyloidosis in China. Kidney Dis (Basel). 2016 Apr;2(1):1-9. doi: 10.1159/000444287. Epub 2016 Feb 25. PMID 27536686
- [Background] Merlini G, Bellotti V. Molecular mechanisms of amyloidosis. N Engl J Med. 2003 Aug 7;349(6):583-96. doi: 10.1056/NEJMra023144. No abstract available. PMID 12904524
- [Background] Wechalekar AD, Gillmore JD, Hawkins PN. Systemic amyloidosis. Lancet. 2016 Jun 25;387(10038):2641-2654. doi: 10.1016/S0140-6736(15)01274-X. Epub 2015 Dec 21. PMID 26719234
- [Background] Perfetto F, Moggi-Pignone A, Livi R, Tempestini A, Bergesio F, Matucci-Cerinic M. Systemic amyloidosis: a challenge for the rheumatologist. Nat Rev Rheumatol. 2010 Jul;6(7):417-29. doi: 10.1038/nrrheum.2010.84. Epub 2010 Jun 8. PMID 20531382
- [Background] Gertz MA. Immunoglobulin light chain amyloidosis: 2016 update on diagnosis, prognosis, and treatment. Am J Hematol. 2016 Sep;91(9):947-56. doi: 10.1002/ajh.24433. PMID 27527836
- [Background] Dingli D, Tan TS, Kumar SK, Buadi FK, Dispenzieri A, Hayman SR, Lacy MQ, Gastineau DA, Hogan WJ, Gertz MA. Stem cell transplantation in patients with autonomic neuropathy due to primary (AL) amyloidosis. Neurology. 2010 Mar 16;74(11):913-8. doi: 10.1212/WNL.0b013e3181d55f4d. PMID 20231668
- [Background] Kumar S, Dispenzieri A, Lacy MQ, Hayman SR, Buadi FK, Colby C, Laumann K, Zeldenrust SR, Leung N, Dingli D, Greipp PR, Lust JA, Russell SJ, Kyle RA, Rajkumar SV, Gertz MA. Revised prognostic staging system for light chain amyloidosis incorporating cardiac biomarkers and serum free light chain measurements. J Clin Oncol. 2012 Mar 20;30(9):989-95. doi: 10.1200/JCO.2011.38.5724. Epub 2012 Feb 13. PMID 22331953
- [Background] Palladini G, Hegenbart U, Milani P, Kimmich C, Foli A, Ho AD, Vidus Rosin M, Albertini R, Moratti R, Merlini G, Schonland S. A staging system for renal outcome and early markers of renal response to chemotherapy in AL amyloidosis. Blood. 2014 Oct 9;124(15):2325-32. doi: 10.1182/blood-2014-04-570010. Epub 2014 Aug 12. PMID 25115890
- [Background] Palladini G, Perfetti V, Obici L, Caccialanza R, Semino A, Adami F, Cavallero G, Rustichelli R, Virga G, Merlini G. Association of melphalan and high-dose dexamethasone is effective and well tolerated in patients with AL (primary) amyloidosis who are ineligible for stem cell transplantation. Blood. 2004 Apr 15;103(8):2936-8. doi: 10.1182/blood-2003-08-2788. Epub 2003 Dec 18. PMID 15070667
- [Background] Jaccard A, Moreau P, Leblond V, Leleu X, Benboubker L, Hermine O, Recher C, Asli B, Lioure B, Royer B, Jardin F, Bridoux F, Grosbois B, Jaubert J, Piette JC, Ronco P, Quet F, Cogne M, Fermand JP; Myelome Autogreffe (MAG) and Intergroupe Francophone du Myelome (IFM) Intergroup. High-dose melphalan versus melphalan plus dexamethasone for AL amyloidosis. N Engl J Med. 2007 Sep 13;357(11):1083-93. doi: 10.1056/NEJMoa070484. PMID 17855669
- [Background] Kastritis E, Wechalekar AD, Dimopoulos MA, Merlini G, Hawkins PN, Perfetti V, Gillmore JD, Palladini G. Bortezomib with or without dexamethasone in primary systemic (light chain) amyloidosis. J Clin Oncol. 2010 Feb 20;28(6):1031-7. doi: 10.1200/JCO.2009.23.8220. Epub 2010 Jan 19. PMID 20085941
- [Background] Huang X, Wang Q, Chen W, Zeng C, Chen Z, Gong D, Zhang H, Liu Z. Induction therapy with bortezomib and dexamethasone followed by autologous stem cell transplantation versus autologous stem cell transplantation alone in the treatment of renal AL amyloidosis: a randomized controlled trial. BMC Med. 2014 Jan 6;12:2. doi: 10.1186/1741-7015-12-2. PMID 24386911
- [Background] Cavo M, Pantani L, Pezzi A, Petrucci MT, Patriarca F, Di Raimondo F, Marzocchi G, Galli M, Montefusco V, Zamagni E, Gamberi B, Tacchetti P, Brioli A, Palumbo A, Sonneveld P. Bortezomib-thalidomide-dexamethasone (VTD) is superior to bortezomib-cyclophosphamide-dexamethasone (VCD) as induction therapy prior to autologous stem cell transplantation in multiple myeloma. Leukemia. 2015 Dec;29(12):2429-31. doi: 10.1038/leu.2015.274. Epub 2015 Oct 7. No abstract available. PMID 26442610
- [Background] Dispenzieri A, Buadi F, Kumar SK, Reeder CB, Sher T, Lacy MQ, Kyle RA, Mikhael JR, Roy V, Leung N, Grogan M, Kapoor P, Lust JA, Dingli D, Go RS, Hwa YL, Hayman SR, Fonseca R, Ailawadhi S, Bergsagel PL, Chanan-Khan A, Rajkumar SV, Russell SJ, Stewart K, Zeldenrust SR, Gertz MA. Treatment of Immunoglobulin Light Chain Amyloidosis: Mayo Stratification of Myeloma and Risk-Adapted Therapy (mSMART) Consensus Statement. Mayo Clin Proc. 2015 Aug;90(8):1054-81. doi: 10.1016/j.mayocp.2015.06.009. PMID 26250727

DOCUMENTS (1):
  • Study Protocol (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT04612582/Prot_000.pdf